CLINICAL TRIAL: NCT01729247
Title: Study to Evaluate the Impact of FeNO Assessments on Asthma Management Decisions in Subject 7 to 60 Years of Age
Status: Completed | Type: Observational
Sponsor: Aerocrine AB (Industry)
Responsible Party: Sponsor
Other Study IDs: AER-043
Record Dates: First submitted 2012-11-12; First posted 2012-11-20 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FeNO: Participants with asthma will have a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit.
  Interventions: Device: NIOX MINO® Instrument (09-1100)

INTERVENTIONS:
Device: NIOX MINO® Instrument (09-1100)

SUMMARY:
Objective: To evaluate the impact of FeNO assessments on asthma treatment decisions.

Secondary objectives: Evaluate the ability of physicians to correctly assess airway inflammation using standard clinical assessment tools (i.e., prior to FeNO measurement). Estimate the cost consequences of changes in asthma management following FeNO determinations

Number of participants: Approximately 40 to 50 subjects will participate in the study during an (approximately) 8-12 week study enrollment period.

Reference product: NIOX MINO® Instrument (09-1100)

Performance assessments: Fractional Exhaled Nitric Oxide (FeNO) Measurements will be performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011).

Response to Study Physician Questions before (Questions 1, 2, and 3) and after (Question 4) FeNO has been measured and seen by the Physician/Health Care Practitioner.

Safety assessments: The Investigator is responsible for the detection, reporting, and documentation of events meeting the definition of an Adverse Event (AE) and/or Serious Injuries as provided in this clinical investigation plan (CIP) from the time that informed consent has been provided and during the study period

Criteria for evaluation: This is an observational, pilot study and there are currently no plans for a formal statistical analysis. Information gained from this study may be used to design subsequent studies in subjects with asthma. Data collected will be summarized in a clinical study report but will not be subject to formal hypothesis testing

DETAILED DESCRIPTION:
INTRODUCTION

Overview:

The measurement of exhaled nitric oxide (FeNO) is the only clinical test for measuring airway inflammation that can be performed consistently and accurately in clinical practice at the point-of-care. Airway inflammation is now recognized as the central mechanism in the pathogenesis of asthma. The measurement of FeNO with the NIOX MINO® device provides a rapid, noninvasive, and inexpensive tool to assess airway inflammation in inflammatory airway diseases such as asthma. The test is easy to perform and requires minimal training for the operator to conduct the test.

Role of Exhaled Nitric Oxide (FeNO):

FeNO has evolved as a predictive and prognostic biomarker for airway inflammation. Nitric oxide (NO) gas is produced in the epithelial cells of the bronchial wall as an intrinsic part of the inflammatory process.

Measuring the amount of FeNO is useful in the initial assessment of patients with chronic cough or non-specific respiratory symptoms suggestive of asthma, and for the management of patients with established asthma who are receiving corticosteroid treatment.

Intended Use:

NIOX MINO® measures Nitric Oxide (NO) in human breath. Nitric Oxide is frequently increased in inflammatory processes such as asthma. The fractional NO concentration in expired breath (FeNO) can be measured by NIOX MINO® with assurance that such measurements are repeatable and according to guidelines for NO measurement established by the American Thoracic Society.

Rationale for Study:

None of the standard clinical assessment tools provide information regarding underlying airway inflammation, the control of which is central to an effective asthma management strategy. Therefore this study will evaluate the impact of FeNO assessments on asthma treatment decisions in approximately 40-50 subjects 7-60 years of age with asthma. This pilot study will also provide information regarding the ability of physicians to correctly assess airway inflammation using standard clinical assessment tools (i.e., prior to FeNO measurement). Finally, this pilot study will allow the cost consequences of changes in asthma management following FeNO determinations to be estimated.

CLINICAL INVESTIGATION OBJECTIVES The primary objective of this study is to evaluate the impact of FeNO assessments on asthma treatment decisions.

The secondary objectives of this study are to:

* Evaluate the ability of physicians to correctly assess airway inflammation using standard clinical assessment tools (i.e., prior to FeNO measurement).
* Estimate the cost consequences of changes in asthma management following FeNO determinations.

CLINICAL INVESTIGATION PLAN

This is a pilot, observational, single-center, single-visit, outpatient study. Approximately 30 to 50 subjects will participate in the study during an (approximately) 8 to 12 week study enrollment period. Eligible subjects who meet the inclusion/exclusion criteria for this study will be invited to participate. The following documentation and information will be provided by subjects:

* Informed consent
* Demographics
* Smoking history (cigarettes only)
* Usual asthma standard of care assessments
* Asthma control test questionnaire
* Spirometry
* Study physician questions

FeNO: FeNO will be performed and the value will be reviewed and record.

Subject discharge from the study:

Once all information has been collected and all procedures have been performed, the subject will be discharged from the clinic and their study participation will be complete

Medical device:

The NIOX MINO® was initially cleared by the FDA on March 4, 2008 as a new hand-held device for the measurement of exhaled Nitric Oxide, a marker of eosinophilic airway inflammation. The most recent clearance by the FDA was on September 2, 2010 for Instrument (09-1100), which will be used in this study. NIOX MINO® can be used in children 7-17 years of age and in adults 18 years of age or older in the initial assessment and management of asthma.

The NIOX MINO® is a 10 second test based on exhaled breath measured at a 50 ml/second flow rate. Results are provided at the point of care within 2 minutes after the successful completion of the breath test. The test cannot be influenced by patient effort or variations in the clinician's test technique.

Definitions:

Adverse event: Any incident where the use of a medical device (including in vitro diagnostics) is suspected to have resulted in an adverse outcome in a patient.

Serious Injury means injury or illness that:

* Is life-threatening
* Results in permanent impairment of a body function or permanent damage to a body structure, or
* Necessitates medical or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure.

Malfunction: the failure of a device to meet its performance specifications or otherwise perform as intended.

Caused or contributed: the death or serious injury was or may have been attributed to a medical device, or that the medical device was or may have been a factor in a death or serious injury, including events occurring as a result of:

* Failure
* Malfunction
* Improper or inadequate design
* Manufacture
* Labeling
* User error

ELIGIBILITY:
Inclusion Criteria:

* Age: 7 to 60 years of age, inclusive
* Sex: Males and Females
* Diagnosis: Asthma

Exclusion Criteria:

* Concurrent Conditions or Disease: Subjects with an established diagnosis of chronic, obstructive pulmonary disease (COPD) cystic fibrosis (CF), bronchiectasis, obliterative bronchiolitis, ciliary dyskinesia, post-viral bronchial hyperresponsive syndrome, or vocal cord dysfunction are excluded from participation
* Cigarette Smoking: Subjects with greater than a 10 pack-year history of cigarette smoking are excluded from participation
* Study Participation Outside of This Protocol: Subjects currently enrolled in studies of Investigational or Non-Investigational Drugs or Medical Devices and/or who participated in these studies within 30 days prior to this study are excluded from participation

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female subjects, 7 to 60 years of age, inclusive, with asthma will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- North Carolina Clinical Research, Raleigh, North Carolina, United States

REFERENCES:
- [Derived] LaForce C, Brooks E, Herje N, Dorinsky P, Rickard K. Impact of exhaled nitric oxide measurements on treatment decisions in an asthma specialty clinic. Ann Allergy Asthma Immunol. 2014 Dec;113(6):619-23. doi: 10.1016/j.anai.2014.06.013. Epub 2014 Jul 22. PMID 25060819

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants expressing interest who met inclusion and exclusion criteria were asked to sign written informed consent prior to participation.
Period: Overall Study
Arm/Group | FeNO
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FeNO
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (15.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 50
Smoking Status [Number; unit: participants] — At study visit, participants responded to a questionnaire regarding their smoking history. Participants were classified as having never smoked, current smoker, or past smoker.
  participants
    Never Smoked | 35
    Current Smoker | 0
    Past Smoker | 15
Current Medications used for Pulmonary and/or Allergy Conditions [Number; unit: participants] — Provided is a summary of medications taken by >= 5% of participants that are used for pulmonary and/or allergy conditions. The most common medications included short-acting beta-agonist bronchodilators (SABA), inhaled corticosteroid (ICS) and long-acting beta-agonist bronchodilators (LABA) combination products, H1-receptor antagonist and ICS
  participants
    SABA | 47
    ICS/LABA Combination | 20
    H1-Receptor Antagonist | 17
    ICS | 10
    Antihistamine | 9
    Intranasal Corticosteroid | 9
    Leukotriene Receptor Antagonist | 8
    Nasal Decongestant | 4

OUTCOME MEASURES:

1. Primary Outcome: FeNO Values by ACT Score
Description: Scores on an asthma control test (ACT) of <=19 indicates less well controlled asthma, scores >19 indicate well controlled asthma. Force exhaled nitric oxide (FeNO) was measured using a NIOX MINO device. FeNO measures were compared against ACT scores.
Time Frame: Study Visit (single visit study). Approximately 1 hour.
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Groups:
- Low ACT Score: Participants who had an asthma control test (ACT) score of <=19, which indicates less well-controlled asthma
- High ACT Score: Participants who had an asthma control test (ACT) score of >19, which indicates well-controlled asthma
Arm/Group | Low ACT Score | High ACT Score
Number analyzed (Participants) | 29 | 21
parts per billion (ppb) | 40.3 (50.84) | 26.3 (21.42)

2. Primary Outcome: FeNO Categorical Levels by ICS Use
Description: Fractional exhaled nitric oxide (FeNO) is measured using a NIOX MINO device. FeNO measurements were categorized into low (<25 ppb), intermediate (>=25 to <=50 ppb) and high (>50 ppb). Number of participants falling into FeNO categories were then categorized as those that used inhaled corticosteroids (ICS) or ICS/long-acting beta-agonist (LABA) and those who did not use ICS or ICS/LABA.
Time Frame: Study visit (single visit study). Approximately1 hour.
Measure: Number; unit: participants
Groups:
- ICS Use: Participants that used inhaled corticosteroids (ICS) or ICS/long-acting beta-agonist (LABA)
- No ICS Use: Participants that did not use inhaled corticosteroids (ICS) or ICS/long-acting beta-agonist (LABA)
Arm/Group | ICS Use | No ICS Use
Number analyzed (Participants) | 29 | 21
participants
  Low FeNO | 18 | 11
  Intermediate FeNO | 6 | 4
  High FeNO | 5 | 6

3. Secondary Outcome: Physician Assessment of Airway Inflammation
Description: Assessment of airway inflammation was performed by an allergist or nurse practitioner/physicians assistant prior to knowledge of forced exhaled nitric oxide (FeNO) results. Airway inflammation was categorized as low, intermediate or high. Mean FeNO results were summarized by the physicians assessment of airway inflammation (low, intermediate, high, or unsure).
Time Frame: Study visit (single visit study) approximately 1 hour
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Groups:
- Low Airway Inflammation; Intermediate Airway Inflammation; High Airway Inflammation: As categorized by physician assessment
Arm/Group | Low Airway Inflammation | Intermediate Airway Inflammation | High Airway Inflammation
Number analyzed (Participants) | 34 | 14 | 2
parts per billion (ppb) | 31.4 (38.16) | 40.6 (51.37) | 42.0 (25.46)

4. Secondary Outcome: Number of Participants Correctly Categorized by True Level of Airway Inflammation
Description: Assessment of airway inflamation was performed by an allergist or nurse practioner/physicians assistant prior to knowledge of forced exhaled nitric oxide (FeNO) results. Airway inflamation was categorized as low, intermediate or high. A summary of the number of participants with correctly identified airway inflammation assessments by the physician for each true level of inflammation are displayed below.
Time Frame: Study visit (single visit study) approximately 1 hour.
Measure: Number; unit: participants correctly categorized
Arm/Group | Low Airway Inflammation | Intermediate Airway Inflammation | High Airway Inflammation
Number analyzed (Participants) | 29 | 10 | 11
participants correctly categorized | 21 | 3 | 1

5. Secondary Outcome: Asthma Management Changes After FeNO Results Were Considered
Description: Assessment of airway inflammation was performed by an allergist or nurse practitioner/physicians assistant prior to knowledge of fractional exhaled nitric oxide (FeNO) results. Airway inflammation was categorized as low, intermediate or high. Based on these assessments asthma medications were prescribed (prior to knowledge of FeNO results). Following the initial prescriptions, the physicians were informed of FeNO results, and any changes to asthma medication prescriptions were recorded. Asthma medications included short-acting beta-agonist (SABA), inhaled corticosteroid (ICS), ICS/long-acting beta-agonist (LABA), leukotriene receptor antagonist (LTRA), and oral corticosteroid (OCS).
Time Frame: Study visit (single visit study). Approximately1 hour.
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 50
participants
  No Changes | 32
  Changes to SABA | 9
  Changes to ICS | 8
  Changes to ICS/LABA Combination | 6
  Changes to LTRA | 2

ADVERSE EVENTS:
Time Frame: Study Visit (single visit study). Approximately 1 hour.
Arm/Group | FeNO
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No